CLINICAL TRIAL: NCT06305494
Title: Genitourinary Syndrome of Menopause in Thai Gynecologic Cancer Survivors: A Cross-sectional Study
Brief Title: Genitourinary Syndrome of Menopause in Thai Gynecologic Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Apiwat Jongjakapun, Principal Investigator, Khon Kaen University
Other Study IDs: HE671008
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Atrophic Vaginitis; Gynecologic Cancer; Lower Urinary Tract Symptoms
Keywords: Genitourinary syndrome of menopause; Gynecologic cancer
MeSH Terms: conditions — Atrophic Vaginitis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women often face common cancers like ovarian, uterine, and cervical cancers. Improvements in cancer detection and treatment mean more women survive. However, survivors can encounter challenges like ongoing pain, treatment complications, and fertility issues.

Treating these cancers often involves surgeries that might include removing ovaries or using pelvic radiation. This can trigger menopause in younger women, causing problems like vaginal dryness, itching, and urinary issues.

Women who've gone through menopause often deal with these symptoms, affecting their daily lives, confidence, and intimate relationships. Though treatments are available, lack of awareness, embarrassment, and not discussing these issues with doctors can make managing them difficult.

The main treatment for these symptoms is using vaginal estrogen, but it might not be suitable for some cancer survivors. Non-hormonal options like lubricants and moisturizers are alternatives. This study in Thailand aiming to explore how common these issues are among gynecological cancer survivors, their feelings about it, and how it affects their quality of life.

DETAILED DESCRIPTION:
Gynecological cancers, encompassing ovarian, endometrial, and cervical cancers, stand as significant health concerns for women. In 2017, a total of 12,354 new cases were diagnosed in Thailand, underlining the prevalence and impact of these conditions. Advances in cancer screening and treatment have notably improved outcomes, resulting in a growing number of survivors. By 2016, the United States alone recorded 15.5 million cancer survivors, with projections indicating a surge to 26.1 million by 2040. However, even with increased survival rates, challenges persist for survivors, encompassing chronic pain, complications from treatment, and disruptions to fertility, menopause, sexual function, and cognitive health.

The treatment landscape for gynecological cancers is diverse, with the general principle for ovarian and endometrial cancers involving surgical staging. This comprehensive approach includes the removal of the uterus, fallopian tubes, both ovaries, peritoneum, pelvic lymph nodes, and any visible lesions. For cervical cancer, treatment varies based on disease stage. Early-stage cases often undergo surgery, potentially followed by pelvic irradiation. In advanced-stage cervical cancer, a combination of pelvic radiation and chemotherapy is commonly employed. In summary, many gynecological cancer treatments involve the removal of both ovaries or pelvic irradiation, inducing menopause in reproductive-age women.

The female lower reproductive system, including the lower urinary tract, is intricately responsive to estrogenic stimulation. When estrogen is lacking, structural changes occur, giving rise to a cluster of symptoms collectively termed the genitourinary syndrome of menopause (GSM). Estrogen deficiency results in thinning of the vaginal epithelium lining, diminished collagen and elastin fibers, reduced blood supply, and moisture decline. These changes manifest as vaginal symptoms, including burning, itching, and pain during intercourse.

Similarly, the urinary tract, deprived of estrogenic stimulation, undergoes alterations such as urethral shortening, thinning of the urethral epithelium, weakened urethral sphincter contractions, and reduced elasticity of the urinary bladder. This cascade of changes results in lower urinary tract symptoms, comprising dysuria, urinary urgency, incontinence, frequency, nocturia, and recurrent urinary tract infections.

Postmenopausal women commonly experience these symptoms, and systematic literature reviews reveal a prevalence ranging from 13 to 87%. Furthermore, the chronic nature of these symptoms tends to intensify over time. Women who undergo early bilateral oophorectomy are more likely to enter menopause sooner, increasing the risk of developing various urogenital symptoms at a younger age.

The impact of these symptoms on women's lives is profound, affecting daily activities, self-confidence, and intimate relationships. Vaginal symptoms, in particular, can lead to sexual dysfunction, exacerbating challenges in family relationships. Concurrently, urinary symptoms contribute to decreased quality of life, with frequency, nocturia, and urgency correlating with the risk of falls and bone fractures. Additionally, these symptoms are associated with depressed mood, anxiety, and embarrassment, further disrupting aspects of life such as sleep, daily commute, social interactions, and sexual relationships.

Despite the significant impact on quality of life, the effective management of vaginal and genitourinary symptoms is impeded by various factors. These include a lack of knowledge and understanding of the diseases and available treatment options, feelings of embarrassment, and the notable observation that medical personnel often fail to inquire about these specific issues during patient consultations.

The primary treatment for genitourinary symptoms is typically the use of vaginal estrogen. However, certain gynecological cancers, such as leiomyosarcoma, endometrial stromal sarcoma, and specific ovarian cancers, preclude the use of estrogen therapy. In such cases, non-hormonal alternatives like vaginal lubricants, moisturizers, and energy-based devices come into consideration.

This study aim to explore the prevalence of GSM among gynecological cancer survivors. The investigation extends to understanding the magnitude of the problem, examining women's attitudes towards the condition, and assessing its broader impact on their quality of life. This comprehensive exploration seeks to contribute valuable insights to the understanding and management of the complex challenges faced by gynecological cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Participant with gynecologic cancer (cancer of ovary, fallopian tube, uterus, cervix, vagina, and vulva.)
* Time passed more than 6 months since last cancer treatment.

Exclusion Criteria:

* Participant not entering menopause after cancer treatment.
* Participant with cancer progression.
* Participant currently suffer from severe pain, fatigue, or discomfort.
* Participant deny to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gynecologic cancer survivors, age more than 18 years old that came to the Gynecology Clinic at Khon Kaen University Hospital for routine cancer surveillance.
Sampling Method: Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of genitourinary syndrome of menopause | Baseline
  Prevalence of genitourinary syndrome of menopause among gynecologic cancer survivor (percent)

SECONDARY OUTCOMES:
Severity of genitourinary syndrome of menopause | Baseline
  Severity of genitourinary syndrome of menopause measured using visual analog scale (range 0-10; 0 is the least severe, 10 is the most severe)
Quality of life of gynecologic cancer survivor | Baseline
  Quality of life score measured using a visual analog scale (range 0-10; 0 is the least negative effect on quality of life, 10 is the most negative effect on quality of life)
Attitude toward genitourinary syndrome of menopause in gynecologic cancer survivor | Baseline
  Assessment of attitude toward genitourinary syndrome of menopause by asking whether participant agreed with the statement or not (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Apiwat Jongjakapun, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No